CLINICAL TRIAL: NCT00397306
Title: Study for the Evaluation of a Bioimpedance Method for Determination of Dry Weight in Dialysis Patients
Brief Title: Evaluation of a Bioimpedance Method for Determination of Dry Weight in Dialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Saarland (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 95/06
Record Dates: First submitted 2006-11-07; First posted 2006-11-09 (Estimated); Last update posted 2009-04-08 (Estimated); Status verified 2009-04

CONDITIONS: Renal Insufficiency, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Bioimpedance Analysis

SUMMARY:
The purpose of this study is the evaluation of a bioimpedance method for determination of dry weight in dialysis patients. Additionally normal tissue hydration in non-Dialysis patients is investigated in healthy subjects and patients with chronic kidney disease in stages K/DIGO I-IV

ELIGIBILITY:
Inclusion Criteria:

* clinically stable on dialysis within the last three months
* signed written informed consent

Exclusion Criteria:

* acute myocardial infarction or stroke within the last six months
* heart failure stage NYHA IV
* concommitant participation in other interventional trials
* psychiatric conditions that prevent subject from following the study procedures / protocol
* pregnancy or lactation
* limb amputation
* cardiac pacemaker
* joint implants
* implantable pumps and other metallic implants

For healthy subjects and CKD patients in stages K/DIGO I-IV the above mentioned criteria other than the first mentioned are applicable respectively.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-11; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Bioimpedance Dry weight

SECONDARY OUTCOMES:
Resistance
Resistivity
Blood pressure
LV Diameter
Shortening Fraction
Wall thickness LA, LV
Quality of Life
EPO-Dose

CONTACTS AND LOCATIONS:
Overall Officials: Eric Seibert, M.D., Principal Investigator — University Hospital of Saarland, Department of Internal Medicine IV, Division of Nephrology and Hypertension
Locations (1):
- University Hospital of Saarland, Dept. of Internal Medicine IV, Div. of Nephrology and Hypertension, Homburg, Saarland, Germany